CLINICAL TRIAL: NCT02210208
Title: An Open, Non-controlled, Multi-centre, Clinical Investigation to Verify Performance and Safety of a Soft Silicone Wound Contact Layer Containing Silver in the Treatment of Skin Grafts in Surgical Burn Patients and the Usefulness of a Marketed Donor Site Dressing.
Brief Title: A Soft Silicone Wound Contact Layer Containing Silver in the Treatment of Skin Grafts in Surgical Burn Patients.
Acronym: MpTAg03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MpTAg03
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Burn Injury; Skin Graft
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Two Parts (part A and B) with one dressing device for the skin graft placed on a surgical burn wound and another dressing device placed on the donor site.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepitel® Ag (Experimental): A dressing device used for surgical burn wounds with skin graft.
  Interventions: Device: Mepitel® Ag
- Mepilex® Transfer Ag (Experimental): Donor site dressing device in the very same patient.
  Interventions: Device: Mepilex® Transfer Ag

INTERVENTIONS:
Device: Mepitel® Ag — A soft silicone wound contact layer that allows exudates to pass vertically into a secondary absorbent dressing. The product provides fixation and protection of the tissues and has antimicrobial properties.
  This silicone net dressing will be used to prevent lifting and adherence of skin grafts to the dressings, as well as to prevent pain, and promote healing.
  Arms: Mepitel® Ag
Device: Mepilex® Transfer Ag — Mepilex® Transfer Ag is a soft silicone wound contact layer that absorbs and transfers exudate, maintains a moist wound healing environment and has antimicrobial properties.
  Mepilex® Transfer Ag consists of a Safetac® adhesive layer and compressed polyurethane foam containing silver sulphate and activated carbon. Safetac® is a unique adhesive technology that minimizes pain to patients and trauma to wounds and the surrounding skin. It minimizes risk for maceration by sealing the wound margins; ensuring exudate does not spread to the surrounding skin.
  Arms: Mepilex® Transfer Ag

SUMMARY:
Part A The primary objective of Part A will be to verify performance and safety of Mepitel® Ag, a meshed, non- adherent soft silicone wound contact layer containing silver in the treatment of skin grafts in surgical burn patients.

Part B The primary objective of Part B will be to examine the usefulness of Mepilex® Transfer Ag as an adequate option for donor site healing.

DETAILED DESCRIPTION:
This post market clinical follow-up investigation is designed as an open, non-controlled, multi- centre, clinical investigation.

A total of approximately 25 subjects from among 4-6 clinical investigative sites will be evaluated providing they fulfill all the inclusion criteria and none of the exclusion criteria. A signed and dated informed consent/assent will be obtained for all subjects.

Subjects to be included will present with a thermal burn injury that will require skin grafting and result in a donor site. Overall percent Total Body Surface Area (%TBSA) burned will not exceed 30%.

The subjects will be consecutively allocated to a subject code providing they fulfill all inclusion criteria and none of the exclusion criteria and have signed a written consent.

The subjects were participating in the study for 14 days postop.

ELIGIBILITY:
Part A

Inclusion Criteria

* Subjects with burn injury resulting in up to 30% TBSA
* Full thickness area of burn should not be more than 20%
* Area in need of skin grafting can be 1-15% TBSA
* Study site area must have healthy, intact peri-wound skin surrounding it to allow for adequate overlap of study product
* Thermal injuries only
* Subjects age 18 months to < 65 years.
* Signed informed consent
* Subjects who are younger than the legal consenting age must in addition to their own assent form have a signature from a legally authorized representative.

Exclusion Criteria

* Greater than 30% TBSA
* Full thickness areas greater than 20% TBSA
* Full thickness area to be grafted less than 1%
* Presence of respiratory involvement
* Subjects on mechanical ventilation
* Subjects with infected burn wounds
* Subjects with organ failure
* Diagnosed underlying disease(s) (e.g. HIV/AIDS, cancer and severe aeaemia) judged by the investigator to be a potential interference in the treatment
* Subjects treated with systemic glucocorticosteroids, except patients taking occasional doses or doses less than 10mg prednisolone/day or equivalent
* Known allergy/hypersensitivity to any of the components of the investigation products.
* Subjects with physical and/or mental conditions that are not expected to comply with the investigation, including patients totally confined to bed
* Participation in other clinical investigation(s) within 1 month prior to start of the investigation
* Previous randomized to this investigation

Part B

Inclusion Criteria

-There must be healthy, intact peri-wound skin surrounding the planned donor site to allow for adequate overlap of study product (5 cm)

Exclusion Criteria

* Investigator do not agree to treat the donor site with Mepilex Transfer Ag
* The subject do not agree to participate in the donor site part

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Glat, Professor, Principal Investigator — Drexel University College of Medicine
Locations (4):
- United States (4):
  - The Arizona Burn Center, Phoenix, Arizona
  - The University of South Florida Board of Trustees, Orlando, Florida
  - Long Island Plastic Surgical Group, New York, New York
  - St. Chrisopher's Hospital for Children, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Mepitel® Ag treatment on graft covered wounds 25 patients. Mepilex® Transfer Ag treatment on donor site 19 patients
Period: Period A (Graft Site)
Arm/Group | Overall Study
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician decided not to graft at OR | 1
Period: Period B (Donor Site)
Arm/Group | Overall Study
Started | 19 (6 subjects was decided by the Physician not to be included in the Part B.)
Completed | 12
Not Completed | 7
Not completed — 7 subjects healed at or before Day 14 | 7

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- All Participants: All participants were enrolled into part A where the subjects were treated with Mepitel Ag on a surgical burn wound. Then, eligible subjects from part A, had skin from a "Donor site" to help the burn wound heal. The "Donor site" was also treated and these patients were included i part B.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] — Population: Participants in Part A=25 and Participants in Part B=19. Every patient in Part A was not eligible for Part B.
  years
    Part A | 28.6 [1 to 62]
    Part B: number analyzed (Participants) | 19
    Part B | 26.9 [3 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All participants were enrolled into part A where the subjects were treated with Mepitel Ag on a surgical burn wound. Then, eligible subjects from part A, had skin from a "Donor site" to help the burn wound heal. The "Donor site" was also treated and these patients were included i part B.
  Participants
    Part A: Female | 6
    Part A: Male | 19
    Part B: number analyzed (Participants) | 19
    Part B: Female | 4
    Part B: Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Healing
Description: Part A: Adequate take of skin graft (defined as at least 95% adherent and healed as assessed by clinical investigator).
Time Frame: 14 days
Population: ITT population. During the surgery, the Phycisian decided that one patient should not receive any skin graft. Therefore there are only 24 patients in Part A and 18 patients in Part B. At Baseline there were 25 ITT patients evaluated for Part A and 19 patients for Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Mepitel Ag: Mepitel Ag treatment on burn wounds with skin grafts
  Mepitel Ag
Arm/Group | Part A: Mepitel Ag
Number analyzed (Participants) | 24
Participants
  Day 7: Graft take healed ≥95%=No | 3
  Day 7: Graft take healed ≥95%=Yes | 21
  Day 14: Graft take healed ≥95%=No | 2
  Day 14: Graft take healed ≥95%=Yes | 22

2. Primary Outcome: Part B
Description: Part B: The healing percentage of donor sites (defined as greater than 95% epithelialization, verified by quantitative photographic analysis).
Time Frame: 14 days with 2 visits
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Mepilex Transfer Ag: Mepilex Transfer Ag treatment at donor site for skin graft.
Arm/Group | Part B: Mepilex Transfer Ag
Number analyzed (Participants) | 18
Participants
  Day 7: Donor site healed ≥95%=No | 15
  Day 7: Donor site healed ≥95%=Yes | 3
  Day 14: Graft take/Donor site healed ≥95%=No: number analyzed (Participants) | 6
  Day 14: Graft take/Donor site healed ≥95%=No | 2
  Day 14: Donor site healed ≥95%=Yes: number analyzed (Participants) | 6
  Day 14: Donor site healed ≥95%=Yes | 4

3. Secondary Outcome: Part A Secondary Outcome.
Description: Satisfactory fixation of the product over the skin graft was assessed by a series of questions regarding the product assessment of product in place at each visit.
  Ability to pass exudate to the secondary dressing was demonstrated by a series of questions regarding the exudate at each visit as well as the adherence of the dressing at removal which would show the ability of the dressing to pass the exudate to the secondary dressing rather than creating eschar between the wound and the dressing.
Time Frame: 14 days with 2 visits
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Mepitel Ag: Mepitel Ag treatment on skin graft over surgical burn wounds.
Arm/Group | Mepitel Ag
Number analyzed (Participants) | 24
Participants
  Day 7: Was a product removal performed: Yes | 24
  Day 7: Was there any adherence to the graft: No | 20
  Day 7: Was there any adherence to the graft: Yes | 4
  Day 7: Graft lift off with removal of product: No | 22
  Day 7: Graft lift off with removal of product: Yes | 2
  Day 14: Was there any adherence to the graft: No | 16
  Day 14: Was there any adherence to the graft: Yes | 3

4. Secondary Outcome: Part B Secondary Outcome.
Description: Ability of Mepilex® Transfer Ag to adhere to donor site without slippage.
Time Frame: 14 days with 2 visits
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Mepilex Transfer Ag
Number analyzed (Participants) | 18
Participants
  Day 7: Was adherence of product assessed: No | 2
  Day 7: Was adherence of product assessed: Yes | 16
  Day 7: Was removal assessment performed: Yes | 3
  Day 7: Did product stick to donor site: No: number analyzed (Participants) | 3
  Day 7: Did product stick to donor site: No | 2
  Day 7: Did product stick to donor site: Yes: number analyzed (Participants) | 3
  Day 7: Did product stick to donor site: Yes | 1
  Day 14: Was adherence of product assessed: Yes: number analyzed (Participants) | 6
  Day 14: Was adherence of product assessed: Yes | 6
  Day 14: Was removal assessment performed: Yes: number analyzed (Participants) | 6
  Day 14: Was removal assessment performed: Yes | 6
  Day 14: Did product stick to donor site: No: number analyzed (Participants) | 6
  Day 14: Did product stick to donor site: No | 6

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- Overall Study: Mepitel Ag treatment and Mepilex Transfer Ag
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=25)
infection (Infections and infestations) | 1 (1) — suspected infection at graft site
infection (Infections and infestations) | 1 (1) — suspected infection at donor site
leukocytosis (Blood and lymphatic system disorders) | 1 (1) — leukosytosis potential from allografted area of burn
hypocalcemia (Blood and lymphatic system disorders) | 1 (1) — hypocalcemia
hypermagnesemia (Blood and lymphatic system disorders) | 1 (1) — hypermagnesemia
hyperphosphatemia (Blood and lymphatic system disorders) | 1 (1) — hyperphosphatemia
hypertension (Blood and lymphatic system disorders) | 1 (1) — hypertension
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) — muscle spasm
femoral artery IV site infiltrated (Surgical and medical procedures) | 1 (1) — femoral artery IV site infiltrated
high blood pressure (Blood and lymphatic system disorders) | 1 (1) — post-op high blood pressure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days